CLINICAL TRIAL: NCT05512806
Title: A Randomized, 6-period, 6-treatment, Single-Dose, Crossover Study to Assess the Pharmacokinetics of AZD5462 Film-coated Tablet Formulation, to Assess the Relative Bioavailability of AZD5462 Film-coated Tablet Formulation vs Oral Solution, and to Assess the Influence of Food on the Pharmacokinetics of AZD5462 in Healthy Participants
Brief Title: A Bioavailability and Food Effect Study of AZD5462 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D9090C00005
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Healthy Participants
Keywords: Healthy participants; Food effect; Relative bioavailability

STUDY DESIGN:
Masking Description: This is an open-label study due to which blinding is not applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment A (Experimental): Participants will receive Dose A orally as a film-coated tablet.
  Interventions: Drug: AZD5462
- Treatment B (Experimental): Participants will receive Dose A orally as a film-coated tablet.
  Interventions: Drug: AZD5462
- Treatment C (Experimental): Participants will receive Dose B orally as a film-coated tablet.
  Interventions: Drug: AZD5462
- Treatment D (Experimental): Participants will receive Dose B orally as an oral solution.
  Interventions: Drug: AZD5462
- Treatment E (Experimental): Participants will receive Dose C orally as a film-coated tablet.
  Interventions: Drug: AZD5462
- Treatment F (Experimental): Participants will receive Dose C orally as a film-coated tablet.
  Interventions: Drug: AZD5462

INTERVENTIONS:
Drug: AZD5462 — Participants will receive AZD5462 orally.

SUMMARY:
This study will assess the pharmacokinetics of AZD5462 film-coated tablet formulation in healthy participants.

DETAILED DESCRIPTION:
This study will consist of six treatment periods.

A total of 16 healthy male and female participants of non-childbearing potential will be randomized in this study to ensure at least 12 evaluable participants at the end of the last treatment period.

The study will comprise of a Screening Period, six Treatment Periods, and a follow-up phone call:

* A screening period of maximum 28 days.
* Six treatment periods during which participants will be residents at the study center from Day -1 until Day 17.

Each participant will receive 6 treatments.

The following treatments will be given:-

* Treatment A: Dose A of AZD5462 film-coated tablet in a fasted state.
* Treatment B: Dose A of AZD5462 film-coated tablet in a fed state.
* Treatment C: Dose B of AZD5462 film-coated tablet in a fasted state.
* Treatment D: Dose B of AZD5462 oral solution in a fasted state.
* Treatment E: Dose C of AZD5462 film-coated tablet in a fasted state.
* Treatment F: Dose C of AZD5462 film-coated tablet in a fed state.
* A follow-up phone call will take place on Day 21 (± 1 day) to record adverse events (AEs) and concomitant medication.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male and female participants aged 18 to 55 years at screening and admission with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative pregnancy test at screening and on admission to the study center, must not be lactating and must be of non-childbearing potential confirmed at screening by fulfilling one of the following criteria:

  1. Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and Follicle-stimulating hormone (FSH)/Luteinizing hormone (LH) levels in the postmenopausal range.
  2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
* Male participant must adhere to the contraception methods details.
* Have a Body mass index (BMI) between 18 and 32 kg/m2 inclusive and weigh at least 50 kg and no more than 105 kg inclusive at screening.

Exclusion Criteria:

* History of any clinically significant disease or disorder which may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* Any of the below conditions:

  1. Systemic sclerosis.
  2. Moderate to severe valvular disease.
  3. Hypertrophic obstructive cardiomyopathy.
  4. Restrictive cardiomyopathy.
  5. Gilbert's syndrome.
  6. History of vascular or left ventricular aneurysms, or prior dissections.
  7. Any history of joint hypermobility, Marfan's Syndrome, or any connective tissue disorder.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of Investigational medicinal product (IMP).
* Any laboratory values with the following deviations at screening, or admission to the study center:

  1. Total bilirubin > Upper limit of normal (ULN).
  2. Alanine aminotransferase > 1.5 × ULN.
  3. Aspartate aminotransferase > 1.5 × ULN.
  4. Estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73m2, as assessed by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.
  5. White blood cell count < 3.5 k/uL and > ULN.
  6. Hemoglobin < Lower limit of normal (LLN).
* Any clinically significant abnormalities in clinical biochemistry, hematology, or urinalysis results.
* Any clinically significant abnormal findings in vital signs after 5 minutes supine rest, at screening or admission defined as any of the following:

  1. Systolic Blood pressure (BP) < 90 mmHg or ≥ 140 mmHg.
  2. Diastolic BP < 50 mmHg or ≥ 90 mmHg.
  3. Heart rate < 50 bpm or > 90 bpm.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting 12-lead Electrocardiogram (ECG) at screening or admission.

  1. Prolonged QTcF > 450 ms.
  2. Shortened QTcF < 340 ms.
  3. Family history of long QT syndrome.
  4. PR(PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation).
  5. PR(PQ) interval prolongation (> 240 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third-degree AV block, or AV dissociation.
  6. Persistent or intermittent complete BBB. Participants with Intraventricular conduction delay (IVCD) with QRS < 120 ms are acceptable if there is no evidence of eg, ventricular hypertrophy, or pre-excitation.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and Human immunodeficiency virus (HIV) antibody.
* Known or suspected history of drug abuse.
* Has received another new chemical entity within 30 days of the first administration of IMP in this study.
* Plasma donation within 1 month of screening or any blood donation/loss > 500 mL during the 3 months prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5462.
* Current smokers or those who have smoked or used nicotine products within the 3 months prior to screening.
* Positive screen for drugs of abuse, alcohol, or cotinine at screening or on each admission to the study center prior to the first administration of the IMP.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, megadose vitamins, and minerals during the 2 weeks or 5 half-lives of the medication, whichever is longer, prior to the first administration of IMP.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* Excessive intake of caffeine-containing drinks or food.
* Participants who have previously received AZD5462.
* Any ongoing or recent minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Participants who are vegans or have medical dietary restrictions.
* Participants who cannot communicate reliably with the Principal Investigator (PI).
* Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* Clinical signs and symptoms consistent with Coronavirus disease 2019 (COVID-19), or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 to Day 17
  The AUCinf of a film-coated tablet of AZD5462 at 3 dose levels will be assessed.
Area under the plasma concentration-curve from time zero to last quantifiable concentration (AUClast) | Day 1 to Day 17
  The AUClast of a film-coated tablet of AZD5462 at 3 dose levels will be assessed.
Maximum observed plasma (peak) drug concentration [Cmax] | Day 1 to Day 17
  The Cmax of a film-coated tablet of AZD5462 at 3 dose levels will be assessed.
Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 to Day 17
  The effect of a high-fat, high-calorie meal in comparison to fasting conditions on the AUCinf of AZD5462 after a single oral dose at 2 dose levels will be assessed.
Area under the plasma concentration-curve from time zero to last quantifiable concentration (AUClast) | Day 1 to Day 17
  The effect of a high-fat, high-calorie meal in comparison to fasting conditions on the AUClast of AZD5462 after a single oral dose at 2 dose levels will be assessed.
Maximum observed plasma (peak) drug concentration [Cmax] | Day 1 to Day 17
  The effect of a high-fat, high-calorie meal in comparison to fasting conditions on the Cmax of AZD5462 after a single oral dose at 2 dose levels will be assessed.
Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 to Day 17
  The relative bioavailability of the film-coated tablet vs oral solution formulation will be determined by the assessment of AUCinf.
Area under the plasma concentration-curve from time zero to last quantifiable concentration (AUClast) | Day 1 to Day 17
  The relative bioavailability of the film-coated tablet vs oral solution formulation will be determined by the assessment of AUClast.
Maximum observed plasma (peak) drug concentration [Cmax] | Day 1 to Day 17
  The relative bioavailability of the film-coated tablet vs oral solution formulation will be determined by the assessment of Cmax.

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs), and Serious Adverse Events (SAEs) | Until follow-up (Day 21)
  The safety, and tolerability of single doses of AZD5462 in healthy participants will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home